CLINICAL TRIAL: NCT05275985
Title: A Prospective Pilot Study to Explore Performance and Efficacy of 68Ga-FAPI PET/CT in Pancreatic Ductal Carcinoma Patients
Brief Title: 68Ga-FAPI PET/CT in Pancreatic Ductal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-FAPIPDAC
Record Dates: First submitted 2022-02-20; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: PDAC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI PET/CT examination (Experimental): Patients with suspected pancreatic lesions underwent 68Ga-FAPI PET/CT to distinguish benign and malignant lesions, to evaluate the resectability of lesions and to detect distant metastasis. The clinicians decided the treatment methods based on the results of 68Ga-FAPI PET/CT.
  Interventions: Diagnostic Test: 68Ga-FAPI Positron Emission Tomography-Computed Tomography

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI Positron Emission Tomography-Computed Tomography — The patients with suspected pancreatic lesions were included. They underwent 68Ga-FAPI PET/CT to distinguish benign and malignant lesions, to evaluate the resectability of lesions and to detect distant metastasis. The treatment methods were decided according to the results of 68Ga-FAPI PET/CT.

SUMMARY:
Fibroblast activation protein (FAP) is overexpressed in cancer-associated fibroblasts (CAFs), which constitutes a major proportion of cells within the tumor microenvironment, especially in primary pancreatic ductal carcinoma (PDAC). In this prospective study, we aimed to evaluate the performance and value of 68Ga-FAPI-04 PET/CT in the patients with PDAC.

DETAILED DESCRIPTION:
With an incidence rate of 10 cases per 100,000 people per year, cancer of the pancreas is the third most common malignancy of the gastrointestinal tract. The overall survival for patients with pancreatic cancer is very poor, with a 5-year survival of 1% to 4%. Successful therapy depends on early diagnosis. The discrimination between benign and malignancies of the pancreas and the assessment of local resectability and distant metastases of the pancreatic cancer remains challenging with different imaging modalities such as ultrasound (US), endoscopic US (EUS), multidetector row computed tomography (MDCT), magnetic resonance imaging (MRI), and 18F-FDG positron emission tomography (PET). PDAC is characterized by a distinct and exuberant desmoplastic stroma, with stromal components outnumbering the pancreatic cancer cells. In PDAC, more than 90% of the tumour volume consists of cancer-associated fibroblasts (CAF). Fibroblast activation protein (FAP) is highly and selectively expressed in CAFs but is weakly expressed or not detected in normal tissues. The aim of this study was to evaluate the impact of FAPI-PET/CT on the clinical management of patients with suspected pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected pancreatic lesions
2. Signed written consent.

Exclusion Criteria:

1. pregnancy;
2. breastfeeding;
3. any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Standard Uptake Value (SUV） | through study completion, an average of 0.5 year
  Determined and compared the SUV for detected lesions in 68Ga-FAPI
The numbers of patients who been changed the treatment methods | through study completion, an average of 0.5 year
  Determination the patients numbers who been changed the treatment methods after 68Ga-FAPI PET
The numbers of lesions | through study completion, an average of 0.5 year
  Determination the lesions numbers were detected by 68Ga-FAPI
Progression Free Survival (PFS) | through study completion, an average of 1 year
  Determination the progression free survival of included patients
Overall Survival (OS) | through study completion, an average of 2 year
  Determination the overall survival of included patients

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospita, Beijing, Beijing Municipality, China